CLINICAL TRIAL: NCT06589518
Title: A Prospective, Single Center Study to Evaluate the Efficacy and Safety of Tenofovir Alafenamide Conversion in Liver Transplant Patients
Brief Title: To Evaluate the Efficacy and Safety of Tenofovir Alafenamide Conversion in Liver Transplant Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jongman Kim (Other)
Responsible Party: Sponsor-Investigator, Jongman Kim, Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-07-122
Record Dates: First submitted 2024-07-31; First posted 2024-09-19 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Hepatitis B Virus; Liver Transplant; Renal Insufficiency
MeSH Terms: conditions — Hepatitis B; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental(Tenofovir alafenamide) (Experimental): Tenofovir alafenamide is administered once every day with 25mg PO.
  Interventions: Drug: Tenofovir Alafenamide Citrate

INTERVENTIONS:
Drug: Tenofovir Alafenamide Citrate — Tenofovir alafenamide is administered once every day with 25mg PO for 48 weeks.
  Other Names: Vemlia

SUMMARY:
This clinical trial aims to confirm the efficacy and safety of Vemlia® tablets (Tenofovir alafenamide) in liver transplant patients with hepatitis B, focusing on their effects on renal function.

HBV reactivation post-liver transplantation can result in a post-transplant mortality rate of up to 50% within two years, making prophylaxis critical. Currently, a combination therapy of HBIG and nucleotide analogues is commonly used. Among the nucleotide analogues (NA), entecavir (ETV) and tenofovir disoproxil fumarate (TDF) are frequently used as first-line therapies. However, both ETV and TDF have nephrotoxicity, requiring caution in patients with chronic kidney disease. Specifically, 18% of liver transplant patients develop chronic kidney disease due to immunosuppressant use, making the appropriate use of antiviral drugs to preserve renal function crucial.

TAF has been reported through RCTs to be more effective than TDF in preserving renal function and bone density, while showing similar antiviral effects. However, these studies have been conducted exclusively on general chronic liver disease patients. Although multicenter studies have been reported for liver transplant patients, they were retrospective and involved a limited number of patients.

Therefore, the primary objective of this study is to assess the impact of converting to TAF on renal function preservation in liver transplant patients taking antivirals for HBV prophylaxis. The secondary objectives are to evaluate the antiviral effect on HBV, the impact on lipid profiles, and the effectiveness in preserving bone density.

DETAILED DESCRIPTION:
TAF has been reported through RCTs to be more effective than TDF in preserving renal function and bone density, while showing similar antiviral effects. However, these studies have been conducted exclusively on general chronic liver disease patients. Although multicenter studies have been reported for liver transplant patients, they were retrospective and involved a limited number of patients.

Therefore, the primary objective of this study is to assess the impact of converting to TAF on renal function preservation in liver transplant patients taking antivirals for HBV prophylaxis. The secondary objectives are to evaluate the antiviral effect on HBV, the impact on lipid profiles, and the effectiveness in preserving bone density.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 19 years or older.
2. Patients who have maintained stable liver graft function for one year after liver transplantation due to HBV and meet the following conditions:

   ALT < 3 x ULN and AST < 3 x ULN
3. Patients taking antiviral therapy other than TAF for HBV prophylaxis.
4. Patients with a tacrolimus trough level maintained between 3-10 ng/mL.
5. Patients who have voluntarily decided to participate in the clinical trial after fully understanding the detailed explanation of the trial and have provided written consent.

Exclusion Criteria:

1. Patients who have undergone transplantation of organs other than the liver or re-transplantation.
2. Patients who have received BAL system treatment or auxiliary partial orthotopic liver transplantation (APOLT) before the transplantation.
3. Patients with concurrent viral infections (HCV, HIV).
4. Patients taking mTOR inhibitors (e.g., Everolimus (Certican), etc.).
5. Patients with eGFR <30 or those undergoing dialysis.
6. Pregnant or breastfeeding women.
7. Patients or their spouses/partners who do not agree to use medically acceptable and appropriate contraception methods* during the clinical trial period.

   * Appropriate contraception methods: hormonal contraception, intrauterine device (IUC or IUS), tubal ligation, tubal occlusion, hysterectomy, vasectomy, double barrier methods (combined use of male or female condoms with cervical caps, diaphragms, or contraceptive sponges), single barrier methods with spermicide.

     8 . Patients with a history of hypersensitivity to Tenofovir. 9 . Patients with genetic disorders such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.

10. Patients who are deemed unsuitable for participation in the clinical trial by the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The amount of eGFR change | Through study completion, an average of 12months
  The amount of eGFR change at 12months after conversion compared to before TAF conversion

SECONDARY OUTCOMES:
The amount of Creatinine change | an average of 12months
  Creatinine status by 12 months after conversion compared to before TAF conversion
The amount of CKD stage change | an average of 12months
  CKD stage status by 12 months after conversion compared to before TAF conversion
effectiveness | Through study completion, an average of 12months
  HBV recurrence rate
BMD change | an average of 12months
  BMD status by 12 months after conversion compared to before TAF conversion

CONTACTS AND LOCATIONS:
Overall Officials: Jongman Kim, Ph, MD, Principal Investigator — Samsung Medical Center